CLINICAL TRIAL: NCT01081912
Title: A Randomized Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Tolerability and Safety of Hydrocodone Bitartrate Controlled-Release Capsules in Opioid-experienced Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Phase 3 Study of Hydrocodone Bitartrate Controlled-release Capsules in Subjects With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZX002-0801
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2014-03

CONDITIONS: Back Pain Lower Back Chronic
Keywords: chronic pain; back pain
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Sugars; Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocodone Bitartrate Capsules (Active Comparator): Hydrocodone Bitartrate Controlled-Release Capsules
  Interventions: Drug: Hydrocodone bitartrate
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Capsules, no active substance, shells identical to active comparator capsules
  Other Names: Sugar pill
  Arms: Placebo comparator
Drug: Hydrocodone bitartrate — dosage form: capsule
  Strengths 10mg, 20mg, 30mg, 40mg, 50mg
  Arms: Hydrocodone Bitartrate Capsules

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Hydrocodone Bitartrate controlled-release capsules in subjects with chronic low back pain.

DETAILED DESCRIPTION:
A randomized Phase 3, placebo-controlled multi-center study to evaluate the safety, efficacy and tolerability of Hydrocodone Bitartrate controlled-release capsules in subjects with chronic low back pain. Subjects will go through an open-label conversion and titration phase followed by a randomized double-blind treatment phase of Hydrocodone (HC)-Controlled-Release (CR) vs. Placebo. The trial will consist of a Screening Phase (up to 14 days), an open-label Conversion and Titration Phase (up to 6 weeks), a 12-week placebo-controlled Treatment Phase, and a 2-week Follow-Up Phone Call

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of moderate to severe chronic lower back pain (CLBP)
* Subjects must be classified as non-neuropathic, neuropathic, or symptomatic for more than 6 months after lower back pain (LBP) surgery
* Subjects must in the Investigator's opinion qualify for around-the-clock opioid therapy for treatment of their chronic lower back pain (CLBP).
* Subjects must have been taking opioids for at least 5 days/week for the past 4weeks
* Subjects must have an average Clinic Pain Score of ≥ 4 on the 11-point (0-10) numeric rating scale (NRS) as an average for the last 24 hours of Screening
* Subjects, in the opinion of the Investigator, must be considered to be in generally good health other then CLBP at Screening
* Female subjects of childbearing potential must have a negative urine pregnancy test at the Screening Visit, and must consent to use a medically-acceptable method of contraception throughout the entire study period.
* Subjects must voluntarily provide written informed consent.

Exclusion Criteria:

* Any clinically significant condition that would, in the opinion of the Investigator, preclude study participation or interfere with the assessment of pain and other symptoms of CLBP or increase the risk of opioid-related adverse events
* A medical condition that, in the opinion of the Investigator, would compromise the subject's ability to swallow, absorb, metabolize, or excrete the study drug
* A surgical procedure for back pain within 6 months
* A nerve or plexus block, including epidural steroid injections or facet blocks
* A history of chemotherapy or confirmed malignancy within past 2 years
* Any other chronic pain condition other than CLBP that, in the Investigator's opinion, would interfere with the assessment of LBP e.g. fibromyalgia, osteoarthritis, rheumatoid arthritis, migraine headaches requiring opioid treatment
* Uncontrolled blood pressure, i.e., subject has a sitting systolic blood pressure >180 mmHg or <90 mmHg, and/or a sitting diastolic blood pressure >120 mmHg or <50 mmHg at Screening
* A Body Mass Index (BMI) >45 kg/m2
* A Hospital Anxiety and Depression Scale (HADS) Index score of >12 in either depression or anxiety subscales or an established history of major depressive disorder that is poorly controlled with medication
* A clinically significant abnormality in clinical chemistry, hematology or urinalysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Romanko, DPM, Study Director — Zogenix, Inc.
Locations (51):
- United States (51):
  - Arizona Research Center, Phoenix, Arizona
  - Clopton Clinic, Jonesboro, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Neuro-Pain Medical Center, Inc., Fresno, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Interwest Rehabilitation, LLC, Littleton, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Gold Coast Research, Plantation, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Perimeter Institute for Clinical Research, Inc., Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Georgia Clinical Research, Snellville, Georgia
  - Suburban Clinical Research, Chicago, Illinois
  - Destiny Clinical Research, LLC, Evansville, Indiana
  - Integrated Clinical Trials Services, Inc., West Des Moines, Iowa
  - International Clinical Research Institute, Leawood, Kansas
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Clinical Trials Management, Metairie, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - River Cities Clinical Research Center, Shreveport, Louisiana
  - NECCR Internal Medicine & Cardiology Associates, LLC, Fall River, Massachusetts
  - Center for Clinical Trials, Biloxi, Mississippi
  - Research West, LLC, Kalispell, Montana
  - Office of Danka Michaels, MD, Las Vegas, Nevada
  - South Jersey Medical Associates, Blackwood, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Center for Clinical Research LLC, Winston-Salem, North Carolina
  - IVA Research, Cincinnati, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Neuropsychiatric Research Center, Oklahoma City, Oklahoma
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Integrity Clinical Research, LLC, Milan, Tennessee
  - InSite Clinical Research, DeSoto, Texas
  - Clinical Trial Network, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Invisions Consultants, LLC, San Antonio, Texas
  - Clinical Trial Network, Spring, Texas
  - Advanced Research Institute, Ogden, Utah
  - Hypothe Test, LLC, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 510 subjects treated with Hydrocodone Bitartrate Extended Release (HC-ER) capsules in the Conversion/Titration Phase, 208 subjects discontinued early and 151 subjects were randomized into each of the two treatment groups (Maintenance HC-ER Treatment and Placebo Treatment).
Groups:
- Conversion/Titration Phase - Open-Label: Conversion/Titration Phase: Hydrocodone Bitartrate Extended Release capsules twice daily for up to 6 weeks (Open-Label Period)
- Double-Blind Treatment Phase: Treatment Phase: Hydrocodone Bitartrate Controlled-Release Capsules twice daily up to 12 weeks (Double-Blind Period)
  Hydrocodone bitartrate: dosage form: capsule
  Strengths 10mg, 20mg, 30mg, 40mg, 50mg
- Double-Blind Treatment Phase: Placebo Comparator: Placebo: Capsules, no active substance, shells identical to active comparator capsules.
  Placebo capsules twice daily for up to 12 weeks (Double-Blind Period)
Period: Conversion/Titration
Arm/Group | Conversion/Titration Phase - Open-Label | Double-Blind Treatment Phase | Double-Blind Treatment Phase: Placebo Comparator
Started | 510 | 0 | 0
Completed | 302 | 0 | 0
Not Completed | 208 | 0 | 0
Not completed — Adverse Event | 47 | 0 | 0
Not completed — Lack of Efficacy | 17 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Protocol Violation | 67 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 0 | 0
Not completed — Non-Compliance | 47 | 0 | 0
Period: Maintenance Treatment
Arm/Group | Conversion/Titration Phase - Open-Label | Double-Blind Treatment Phase | Double-Blind Treatment Phase: Placebo Comparator
Started | 0 | 151 | 151
Completed | 0 | 124 | 59
Not Completed | 0 | 27 | 92
Not completed — Adverse Event | 0 | 2 | 12
Not completed — Lack of Efficacy | 0 | 14 | 64
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 5 | 5
Not completed — Non-Compliance | 0 | 4 | 7
Not completed — Withdrawal by Medical Monitor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Out of 510 subjects treated with Hydrocodone Bitartrate Extended Release (HC-ER) capsules in the Conversion/Titration Phase, 208 subjects discontinued early and 151 subjects were randomized into each of the two treatment groups (Maintenance HC-ER Treatment and Placebo Treatment).
Groups:
- Open-label Conversion/Titration Phase: Hydrocodone Bitartrate Extended Release capsules twice daily for up to 6 weeks (Open-Label)
Arm/Group | Open-label Conversion/Titration Phase
Number analyzed (Participants) | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 462
  >=65 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273
  Male | 237
Region of Enrollment [Number; unit: participants]
  United States | 510

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in 24-hour Pain Intensity Ratings Scale (NRS).
Description: Change in average pain intensity as measured daily by Numeric Rating Scale (NRS) for Pain (0-10; where 0 = no pain, 10 = worst pain imaginable) comparing HC-ER with Placebo. Lower number equals better outcome.
Time Frame: Baseline to Day 85 (Treatment Phase)
Population: The primary efficacy analysis used the Intent to treat (ITT) population which included all 302 randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hydrocodone Bitartrate Capsules: Hydrocodone Bitartrate Controlled-Release Capsules
  Hydrocodone bitartrate: dosage form: capsule
  Strengths 10mg, 20mg, 30mg, 40mg, 50mg
Arm/Group | Hydrocodone Bitartrate Capsules | Placebo Comparator
Number analyzed (Participants) | 151 | 151
units on a scale | 0.48 (1.563) | 0.96 (1.550)

2. Secondary Outcome: Mean Change of the Clinic NRS Pain Intensity
Description: The change in pain intensity as measured in the clinic by a 0-10 Numeric Rating Scale (NRS)
Time Frame: Baseline to Day 85 visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded up to 19 weeks, beginning at the Conversion and Titration Phase through 14 days after the last treatment administration (Treatment Phase).
Description: Subjects received a follow-up phone call 14 days after the end of study (day 85 or early termination) to collect information regarding ongoing AEs or new serious AEs that occurred during this time.
Groups:
- Open-Label Conversion/Titration Phase: Hydrocodone Bitartrate Extended Release capsules twice daily for up to 6 weeks (Open-Label Period)
- Double Blind Treatment Phase: Hydrocodone Bitartrate Capsules: Hydrocodone Bitartrate Controlled-Release Capsules twice daily up to 12 weeks (Double-Blind Period)
  Hydrocodone bitartrate: dosage form: capsule
  Strengths 10mg, 20mg, 30mg, 40mg, 50mg
- Double Blind Treatment Phase: Placebo Comparator: Placebo: Capsules, no active substance, shells identical to active comparator capsules.
  Placebo capsules twice daily for up to 12 weeks (Double-Blind Period)
Arm/Group | Open-Label Conversion/Titration Phase | Double Blind Treatment Phase: Hydrocodone Bitartrate Capsules | Double Blind Treatment Phase: Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 6/510 | 10/151 | 0/151
Other Adverse Events (participants affected / at risk) | 253/510 | 60/151 | 46/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Conversion/Titration Phase (N=510) | Double Blind Treatment Phase: Hydrocodone Bitartrate Capsules (N=151) | Double Blind Treatment Phase: Placebo Comparator (N=151)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Ovarian abscess (Infections and infestations) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Conversion/Titration Phase (N=510) | Double Blind Treatment Phase: Hydrocodone Bitartrate Capsules (N=151) | Double Blind Treatment Phase: Placebo Comparator (N=151)
Constipation (Gastrointestinal disorders) | 56 | 12 | 0
Nausea (Gastrointestinal disorders) | 50 | 11 | 5
Somnolence (Nervous system disorders) | 24 | 1 | 0
Fatigue (General disorders) | 21 | 1 | 2
Headache (Nervous system disorders) | 19 | 0 | 2
Dizziness (Nervous system disorders) | 17 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 16 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 7 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 13 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 8 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 5
Insomnia (Psychiatric disorders) | 12 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 4 | 8
Withdrawal syndrome (Psychiatric disorders) | 3 | 1 | 9
Hypoacusis (Ear and labyrinth disorders) | 3 | 5 | 4
Sinusitis (Infections and infestations) | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days